CLINICAL TRIAL: NCT02940652
Title: Position of Laryngeal Mask in Paediatric Patients During Magnetic Resonance Imaging: Prospective Observational Cohort Study
Brief Title: Laryngeal Mask Position in Magnetic Resonance Imaging in Children
Acronym: LPIMRICH
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, doc.MD.Ph.D, Brno University Hospital
Other Study IDs: KDAR FN Brno 2016
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Laryngeal Mask Malposition
Keywords: Laryngeal mask,MRI
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Paediatric patients undergoing MRI scanning: All paediatric patients undergoing elective MRI scanning of the brain and/or brain and cervical spine
  Interventions: Radiation: Magnetic resonance imaging

INTERVENTIONS:
Radiation: Magnetic resonance imaging — No intervention - description of the position of the LMA obtained during routine elective MRI scanning of the brain and/or cervical spine
  Other Names: MRI

SUMMARY:
The aim of the trial is to obtain and to describe the position of the laryngeal mask during elective magnetic resonance imaging in paediatric patient. The radiologic findings will be compared to the clinical performance of the laryngeal mask.

DETAILED DESCRIPTION:
Properly inserted laryngeal mask (LMA) with good clinical performance can be misplaced (on radiological imaging) but with not know effect on clinical practice. The percentage of the misplaced LMAs are relatively high, but the exact number in paediatric population is currently not clear. The aim of this prospective observational cohort study is to describe the percentage of misplaced LMAs during elective magnetic resonance imaging (MRI) in paediatric patient. After approval of the local ethical committee all elective paediatric patients in study interval (10/2016-3/2017) indicated for elective MRI of the brain or elective MRI of the brain and cervical spine will be included to the trial. Demographic characteristics - age, weight, comorbidities, anesthesia management - education of anesthesiologist, type of LMA, number of insertion attempts, clinical performance of the LMA, presence/absence of leak, the peak inspiratory pressure (mechanical ventilation), volume of air in cuff, complications during anesthesia and LMA soil after extraction - blood, saliva, mucus, gastric content. The clinical performance will be compared to the LMA position on MRI - position of the proximal and the distal site of the LMA cuff according to the cervical vertebrae, displacement of the epiglottis, distance between proximal LMA cuff and vocal cords, distance between distal LMA cuff and vocal cords.

ELIGIBILITY:
Inclusion Criteria:

* paediatric patient undergoing elective MRI scanning - brain and/or brain and cervical spine
* laryngeal mask inserted for airway management during anesthesia
* age between 29 days and 19 years

Exclusion Criteria:

* outside the age limit
* laryngeal mask contraindication - gastroesophageal reflux disease, ileus, full stomach, impairment of the haemodynamics

Ages: 28 Days to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Paediatric patients undergoing elective magnetic resonance imaging of the head (brain) and/or head (brain) and cervical spine
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2016-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Displacement of the laryngeal mask on the MRI imaging | 6 months
  position of the proximal and the distal site of the LMA cuff according to the cervical vertebrae distance between proximal LMA cuff and vocal cords

SECONDARY OUTCOMES:
Clinical performance of the LMA | 6 months
  complications associated with airway management
Demographic characteristics | 6 months
  age, weight, comorbidities

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, doc.MD.Ph.D, Study Director — University Hospital Brno
Locations (1):
- University Hospital Brno, Brno, Jihomoravský Kraj, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Klucka J, Senkyrik J, Skotakova J, Stoudek R, Toukalkova M, Krikava I, Marecek L, Pavlik T, Stouracova A, Stourac P. Laryngeal mask airway Unique position in paediatric patients undergoing magnetic resonance imaging (MRI): prospective observational study. BMC Anesthesiol. 2018 Oct 24;18(1):153. doi: 10.1186/s12871-018-0617-2. PMID 30355285
- See also: Full text open access — https://bmcanesthesiol.biomedcentral.com/articles/10.1186/s12871-018-0617-2